CLINICAL TRIAL: NCT00238706
Title: Left Atrial Radiofrequency Ablation During Mitral Valve Surgery for Continuous Atrial Fibrillation: A Prospective Randomized Clinical Trial
Brief Title: Use of Radiofrequency Ablation to Eliminate Continuous Atrial Fibrillation in Patients Undergoing Mitral Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHF PG/2001096
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-10

CONDITIONS: Atrial Fibrillation; Radiofrequency Catheter Ablation
Keywords: Radiofrequency catheter ablation; Atrial fibrillation; Randomized trial
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency ablation

SUMMARY:
The aim of this prospective randomized clinical trial was to evaluate the early and late outcome following left atrial radiofrequency ablation during MV surgery for the treatment of continuous atrial fibrillation and to assess the functional effects of restoration of sinus rhythm.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a frequent and important contributor to symptoms and morbidity in patients with mitral valve (MV) disease.Radiofrequency ablation (RFA) of the left atrium (LA) during open- heart surgery has emerged as a novel surgical modality for the treatment of AF. Although RFA therapy of the LA is being increasingly offered to patients with chronic AF undergoing MV surgery, its efficacy has not been tested in the context of an adequately powered randomized study. The aim of this prospective randomized clinical trial was to evaluate the early and late outcome following left atrial RFA during MV surgery for the treatment of continuous AF and to assess the functional effects of restoration of SR.

Patients were randomized to undergo MV surgery or MV surgery plus RFA of the LA. Additional cardiac procedures were performed as required.

The primary outcome endpoint was the presence of SR at 12 months. Secondary endpoints included patient functional status and exercise capacity, LA contractility, and LA and left ventricular (LV) dimension and function and plasma levels of B-Type natriuretic peptide (BNP).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring MV surgery with at least 6 month history of atrial fibrillation

Exclusion Criteria:

* Patients with sick sinus syndrome
* Hyperthyroidism
* Permanent pacemaker
* Previous cardiac surgery

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-12; Study Completion 2004-11

PRIMARY OUTCOMES:
The primary outcome endpoint was the presence of SR at 12 months

SECONDARY OUTCOMES:
Secondary endpoints included:
patient functional status and exercise capacity
Left atrial contractility
Left atrial and left ventricular dimension and function Plasma levels of B-Type natriuretic peptide (BNP).

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh Samani, FRCP, Study Director — University of Leicester, Dept of Cardiology

REFERENCES:
- [Result] Doukas G, Samani NJ, Alexiou C, Oc M, Chin DT, Stafford PG, Ng LL, Spyt TJ. Left atrial radiofrequency ablation during mitral valve surgery for continuous atrial fibrillation: a randomized controlled trial. JAMA. 2005 Nov 9;294(18):2323-9. doi: 10.1001/jama.294.18.2323. PMID 16278360